CLINICAL TRIAL: NCT01137370
Title: The Impact of Vitamin D Level and Single Nucleotide Polymorphisms of Vitamin D Receptor Gene on the Development and Treatment Response of Tuberculosis
Brief Title: The Impact of Vitamin D on Tuberculosis Among Koreans
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Joon Yim, Professor, Seoul National University Hospital
Other Study IDs: H-0911-066-301
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-01

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serums for vitamin D measurement DNA for genotyping of vitamin D receptor gene
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with TB
- People without TB

SUMMARY:
Vitamin D has been regarded to be beneficial to tuberculosis (TB) patients. The aim of this study is to elucidate the role of vitamin D deficiency in development and treatment outcomes among Korean TB patients. Furthermore, the impact of genotypes of vitamin D receptor gene on TB development will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* older than 19 years
* diagnosed and treated having a tuberculosis

Exclusion Criteria:

* positive HIV antibody

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed and treated as having a TB in Seoul National University Hospital
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: from April 2010 to March 2011, at Seoul National University Hospital, a tertiary referral hospital in Seoul, South Korea
Pre-assignment Details: Korean who had been abroad for longer than 1 month during the previous year and non-Koreans were excluded from both arms.
Period: Overall Study
Arm/Group | Patients With TB | People Without TB
Started | 116 | 87
Completed | 116 | 87
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With TB | People Without TB | Total
Number analyzed (Participants) | 116 | 87 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 78 | 69 | 147
  >=65 years | 37 | 17 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (18.20) | 50.9 (15.20) | 51.7 (16.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 49 | 101
  Male | 64 | 38 | 102
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 116 | 87 | 203

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Vitamin D Deficiency
Time Frame: At enrollment
Measure: Number; unit: participants, %
Arm/Group | Patients With TB | People Without TB
Number analyzed (Participants) | 116 | 87
participants, % | 36.2 | 27.3

2. Primary Outcome: Median 25-OHD Level
Time Frame: August 2010 to March 2011
Reporting Status: Not Posted, anticipated posting 2011-10
Measure: Number (95% Confidence Interval); unit: participants, ng/mL

ADVERSE EVENTS:
Arm/Group | Patients With TB | People Without TB
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
We did not evaluate the participants' dietary intake of vitamin D or their outdoor activities,and DEXA and PTH were not measured which indicate vitamin D insufficiency.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes